CLINICAL TRIAL: NCT04931160
Title: B-dependant Rare AutoImmune diseaSES - Cohort of Patients With Suspected Diagnosis of Primitive Sjögren Syndrome
Acronym: BRAISES-DiaPSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRAISE DiaPSS
Record Dates: First submitted 2019-12-23; First posted 2021-06-18 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Blood Specimen Collection; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: * Sjögren patients
  * Non-Sjögren controls (retrospective)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sjögren patients (Active Comparator): patients diagnosed Sjögren
  Interventions: Other: Blood, fluid, sells and urine samples
- Non-Sjögren witnesses (Other): patients diagnosed no Sjögren
  Interventions: Other: Blood, fluid, sells and urine samples

INTERVENTIONS:
Other: Blood, fluid, sells and urine samples — Blood, fluid, sells and urine samples will be collected.

SUMMARY:
The objectif is to study the diagnosis performance of the different classification criteria in reference to the gold standard consisting of the diagnosis made by expert doctors after standardized assessment, of pSS (primary Sjogren syndrome)

DETAILED DESCRIPTION:
The formation of this patient is single-center prospective intervention. It consists of collecting data from patients suspected of pSS from standardized biological clinical data and imaging examination and additional pathology.

* Sjögren patients will be followed at inclusion, 2y, 3y, 4y, 6y, 8y and 10 years. Blood, fluid, sells and urine samples will be collected at inclusion, 4y et 10y.
* Non-Sjögren controls will be followed at inclusion and 4y and samples will be collected at the same visits.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Suspicion of SSp (clinical or biological criteria, i.e. dry eye or oral syndrome, arthritis, parotidomegaly, neuropathy, kidney or lung disease...)
* Patient affiliated with Social Security
* Patient who has signed written informed consent

Exclusion Criteria:

* Refusal to participate
* Pregnant and lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2035-02-10 (Estimated); Study Completion 2035-02-10 (Estimated)

PRIMARY OUTCOMES:
Description specificity of different classification criteria FOR sJOGREN (EULAR/ACR 2019, european criteria) | Inclusion
  Specificity of different classification criteria, the standard gold being the diagnosis obtained by consensus of expert doctors after standardized assessment.

SECONDARY OUTCOMES:
Number of patients with different manifestation including in the ESSDAI (Eular Sjögren Syndrome Disease Activity index), gold standard to measure | 10 years
  number of patients wit arthritis of more than 6 joints, parotidomegaly, intertitial lung disease
Number of patients with rheumatological manifestations | 10 years
  number of patients wit arthritis of more than 6 joints, parotidomegaly, intertitial lung disease
Number of patients with dermatological manifestations | 10 years
  number of patients wit arthritis of more than 6 joints, parotidomegaly, intertitial lung disease
Description diagnostic performance of new tests | 10 years
  after evaluation of all différents test performed added to the classical items of the ACR 2017: ie ultrasound parenchymal abnormalities, sub population of B cells....
Disease evolution criteria | 10 years
  modification of the ESSDAI at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Devauchelle, Principal Investigator — CHRU Brest
Locations (1):
- CHRU de Brest, Brest, France